CLINICAL TRIAL: NCT00786591
Title: Clinical Evaluation of Novel Biological Markers for the Prediction of Severe Acute Pancreatitis
Brief Title: Study of New Biological Markers for Prediction of Severe Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Medicine, Professor & Senior Consultant Gastroenterologist, Ho Khek Yu, National University Hospital, Singapore
Other Study IDs: D/05/194
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; biological markers; substance P; hydrogen sulfide; disease severity index
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood; Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute Pancreatitis Patients: Patients presenting with clinical features compatible with acute pancreatitis
- Control: Preoperative patients going for elective cholecystectomy

SUMMARY:
Acute pancreatitis refers to inflammation of the pancreas and is associated with sudden onset of severe abdominal pain, often accompanied by transient systemic manifestations, including fever. In the majority of cases, the inflammatory process is self limiting and patient recovers uneventfully; however, in about 20% to 30% of the cases, a protracted clinical course ensues and the disease may progress to a severe necrotizing form, often triggering a systemic inflammatory response syndrome during which time, acute respiratory distress syndrome, renal failure, shock, and disseminated intravascular coagulation may occur. In the worst sequelae, multiple organ dysfunctions may follow and death supervene. The clinical outcome of patients suffering from severe acute pancreatitis depends to a great extent on the early diagnosis and prediction of severity and timely therapeutic intervention to prevent local and systemic complications. However, the course of the disease is often difficult to predict from the outset. Currently, there is still no single clinical or laboratory test that can be considered the "gold standard" for diagnosis and/or assessment of severity of acute pancreatitis. For a disease that may progress rapidly without apparent sign, the ideal marker for the prediction of disease severity in a patient would be one that is measurable rapidly and easily, besides being able to fulfill all the other criteria required of a good biological marker. To identify such a potential marker for acute pancreatitis requires understanding of the pathophysiological process underlying the rapid progression of a fulminant course of the disease. Although much remains to be elucidated, recent studies in animals have suggested that inflammatory mediators substance P and hydrogen sulfide may play critical roles. This study will evaluate if inflammatory mediators substance P and hydrogen sulfide are upregulated early on in the disease process, and if the levels of their elevation predict disease severity.

ELIGIBILITY:
Inclusion Criteria:

The patient should fulfill all of the following criteria:

* The subject should be at least 18 years of age.
* Clinical features compatible with acute pancreatitis.
* First symptoms of acute pancreatitis not more than 72 hours before enrolment.
* Serum amylase level above 480 U/dl (normal 60-160 U/dl or 2-hour urinary amylase greater than 1120 U (normal 280 U).
* Serum lipase levels greater than 2 U (normal < 1 U).
* Patient has signed consent form regarding participation in the study.

Exclusion Criteria:

The patient should not present any of the following criteria:

* Symptoms of acute pancreatitis present for more than 72 hours
* Clinical evidence of sepsis or other inflammatory diseases.
* Clinical evidence of disorders/disease known to affect endogenous regulation of substance P, e.g. asthma, immune-complex-mediated lung injury, arthritis.
* Age under 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical presentation suggestive of acute pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2006-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Levels of substance P and hydrogen sulfide in blood measured 6-hourly over a time course of 3 days | On admission to hospital, blood sampling will be done every 6 hours for 3 days

SECONDARY OUTCOMES:
Disease severity index derived from: (i) Ranson score; (ii) Acute Physiology and Chronic Health Evaluation (APACHE) II scores; (iv) Glasgow and (v) Multi-Organ System Failure (MOSF) Score | Within 3 days of hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Tamizhselvi R, Moore PK, Bhatia M. Hydrogen sulfide acts as a mediator of inflammation in acute pancreatitis: in vitro studies using isolated mouse pancreatic acinar cells. J Cell Mol Med. 2007 Mar-Apr;11(2):315-26. doi: 10.1111/j.1582-4934.2007.00024.x. PMID 17488480
- [Background] Bhatia M, Zhi L, Zhang H, Ng SW, Moore PK. Role of substance P in hydrogen sulfide-induced pulmonary inflammation in mice. Am J Physiol Lung Cell Mol Physiol. 2006 Nov;291(5):L896-904. doi: 10.1152/ajplung.00053.2006. Epub 2006 Jun 23. PMID 16798781
- [Background] Hegde A, Bhatia M. Neurogenic inflammation in acute pancreatitis. JOP. 2005 Sep 10;6(5):417-21. PMID 16186661
- [Background] Lau HY, Wong FL, Bhatia M. A key role of neurokinin 1 receptors in acute pancreatitis and associated lung injury. Biochem Biophys Res Commun. 2005 Feb 11;327(2):509-15. doi: 10.1016/j.bbrc.2004.12.030. PMID 15629143
- [Background] Grady EF, Yoshimi SK, Maa J, Valeroso D, Vartanian RK, Rahim S, Kim EH, Gerard C, Gerard N, Bunnett NW, Kirkwood KS. Substance P mediates inflammatory oedema in acute pancreatitis via activation of the neurokinin-1 receptor in rats and mice. Br J Pharmacol. 2000 Jun;130(3):505-12. doi: 10.1038/sj.bjp.0703343. PMID 10821777
- [Background] Bhatia M, Saluja AK, Hofbauer B, Frossard JL, Lee HS, Castagliuolo I, Wang CC, Gerard N, Pothoulakis C, Steer ML. Role of substance P and the neurokinin 1 receptor in acute pancreatitis and pancreatitis-associated lung injury. Proc Natl Acad Sci U S A. 1998 Apr 14;95(8):4760-5. doi: 10.1073/pnas.95.8.4760. PMID 9539812